CLINICAL TRIAL: NCT02616926
Title: Hepatic Resection Versus Transarterial Chemoembolization Plus Radiofrequency Ablation for Barcelona Clinic Liver Cancer Stage B Hepatocellular Carcinoma
Brief Title: Hepatic Resection Versus TACE+RFA for BCLC Stage B Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Baogang Peng, Director, Department of Hepatic Surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015012
Record Dates: First submitted 2015-10-25; First posted 2015-11-30 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; hepatectomy; transarterial chemoembolization; radiofrequency ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepatic resection (Experimental): Hepatic resection is performed as a primary treatment for hepatocellular carcinoma.
  Intervention: Hepatic resection
  Interventions: Procedure: Hepatic resection
- TACE + RFA (Active Comparator): TACE is performed as a primary treatment for hepatocellular carcinoma. RFA will be performed two weeks later if necessary.
  Intervention: TACE; RFA
  Interventions: Procedure: TACE; Procedure: RFA

INTERVENTIONS:
Procedure: Hepatic resection — Anatomical surgical resection of the liver including the tumor. Make sure the resection margin is negative during the process.
  Other Names: hepatectomy
  Arms: Hepatic resection
Procedure: TACE — TACE will be performed according to the standard procedure of TACE and will be repeated every four months if needed
  Other Names: transcatheter arterial chemoembolization
  Arms: TACE + RFA
Procedure: RFA — RFA will be performed 1 week after TACE.
  Other Names: radiofrequency ablation
  Arms: TACE + RFA

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common cancer in the world. For patients with intermediate HCC (BCLC stage B), transarterial chemoembolization (TACE) has been recommended as the standard therapy in many clinical practice guidelines. The combination of TACE and radiofrequency ablation (RFA) has also been reported as an effective treatment. However, more and more retrospective studies have reported better therapeutic efficacy of hepatic resection than TACE for intermediate HCC. The purpose of this study was to compare the efficacy of hepatic resection versus TACE+RFA for the treatment of intermediate HCC through prospective randomized clinical trial.

DETAILED DESCRIPTION:
Barcelona Clinic Liver Cancer (BCLC) staging system is the most widely used stage classification for HCC management. For patients with intermediate HCC, palliative treatment transarterial chemoembolization (TACE) was recommended as first choice treatment. However, this recommendation remains controversial. The advice for diagnosis and treatment of HCC from former Chinese Ministry of Health indicated that BCLC may not be suitable in China as most HCC patients were found in intermediate or advanced stage. In recent years, more and more studies declared surgical resection as a better choice for HCC patients in BCLC stage B. However, lack of randomization, small sample size and lack of prospective studies limit the strength of evidence.

To solve this dilemma, a prospective randomized control study was performed to compare the efficacy (1-, 2-, 3-year survival) between surgical resection group and TACE plus radiofrequency ablation group in HCC patients in intermediate stage. This study will provide powerful evidence regarding the better treatment option for HCC patients in BCLC B stage, which will benefit the treatment efficacy of HCC patients in BCLC B stage.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular Carcinoma diagnosed by biopsy or imaging criteria (CT/MRI) and AFP
2. Signed informed consent before registration on study
3. Child-Pugh class A or B
4. Eastern Cooperative Oncology Group Performance status between 0 and 2.
5. BCLC stage B ( diameter of the single tumor ≥5cm or number of tumors ≥3)
6. Hepatitis B history or HBsAg positive
7. Age between 18 and 65 years
8. No previous treatment
9. Laboratory examination test: Platelet count ≥100×109/L; ALT/AST ≤ 3 x ULN; Cr1.5≤ x ULN; INR < 1.5 or PT< ULN +4s; Alb≥30g/L; Tbil≤34mmol/L
10. For patients in Hepatic resection group: radical surgery will be performed: (1) No segmental, lobar or main portal vein and bile duct thrombosis; (2) no lymph nodes metastasis; (3) no extra hepatic metastasis.

Exclusion Criteria:

1. cachexia or poor physical condition;
2. pregnant or HCG positive;
3. Portal vein and bile duct thrombosis or with extra hepatic metastasis.
4. Uncontrolled or refractory ascites or history of hepatic encephalopathy
5. Severe heart, brain or kidney diseases
6. hemophilia or patients with coumarin derivative therapy.
7. .history of organ transplantation or mental disease.
8. Be allergic to adriamycin, lobaplatin, mitomycin or iodized oil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years
  compare 3-year overall survival between the two arms

SECONDARY OUTCOMES:
disease free survival | 3 years
  compare 3-year disease free survival between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Baogang Peng, MD, Principal Investigator — First Affiliated Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - Department of Hepatobiliary Surgery, Cancer Center of Sun-Yat Sen University, Guangzhou, Guangdong
  - Department of Hepatobiliary Surgery, Sun-Yat Sen Memorial Hospital, Guangzhou, Guangdong
  - Department of Hepatic Surgery, First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong

REFERENCES:
- [Result] Torzilli G, Belghiti J, Kokudo N, Takayama T, Capussotti L, Nuzzo G, Vauthey JN, Choti MA, De Santibanes E, Donadon M, Morenghi E, Makuuchi M. A snapshot of the effective indications and results of surgery for hepatocellular carcinoma in tertiary referral centers: is it adherent to the EASL/AASLD recommendations?: an observational study of the HCC East-West study group. Ann Surg. 2013 May;257(5):929-37. doi: 10.1097/SLA.0b013e31828329b8. PMID 23426336
- [Result] Zhong JH, Xiang BD, Gong WF, Ke Y, Mo QG, Ma L, Liu X, Li LQ. Comparison of long-term survival of patients with BCLC stage B hepatocellular carcinoma after liver resection or transarterial chemoembolization. PLoS One. 2013 Jul 9;8(7):e68193. doi: 10.1371/journal.pone.0068193. Print 2013. PMID 23874536
- [Result] Ng KK, Vauthey JN, Pawlik TM, Lauwers GY, Regimbeau JM, Belghiti J, Ikai I, Yamaoka Y, Curley SA, Nagorney DM, Ng IO, Fan ST, Poon RT; International Cooperative Study Group on Hepatocellular Carcinoma. Is hepatic resection for large or multinodular hepatocellular carcinoma justified? Results from a multi-institutional database. Ann Surg Oncol. 2005 May;12(5):364-73. doi: 10.1245/ASO.2005.06.004. Epub 2005 Mar 31. PMID 15915370
- [Result] Peng ZW, Zhang YJ, Chen MS, Xu L, Liang HH, Lin XJ, Guo RP, Zhang YQ, Lau WY. Radiofrequency ablation with or without transcatheter arterial chemoembolization in the treatment of hepatocellular carcinoma: a prospective randomized trial. J Clin Oncol. 2013 Feb 1;31(4):426-32. doi: 10.1200/JCO.2012.42.9936. Epub 2012 Dec 26. PMID 23269991